CLINICAL TRIAL: NCT00000595
Title: Evaluation of Subcutaneous Desferrioxamine as Treatment for Transfusional Hemochromatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Treatment
Other Study IDs: 401
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2000-05

CONDITIONS: Anemia (Iron-Loading); Beta-Thalassemia; Hematologic Diseases; Hemoglobinopathies; Thalassemia; Iron Overload; Hemochromatosis
MeSH Terms: conditions — Anemia; beta-Thalassemia; Hematologic Diseases; Hemoglobinopathies; Thalassemia; Iron Overload; Hemochromatosis | interventions — Deferoxamine

INTERVENTIONS:
Drug: deferoxamine

SUMMARY:
To determine whether deferoxamine prevented the complications of transfusional iron overload.

DETAILED DESCRIPTION:
BACKGROUND:

The prognosis of congenital or long-term anemia was formerly limited by the complications of blood transfusion, splenectomy, or infection, problems now largely overcome by sophisticated clinical care. Lifespan is now determined by the rate of myocardial iron deposition, with death occurring from cardiac failure or arrhythmia, usually between the ages of 15 and 25. Endocrine complications and hepatic enlargement are also evident by this age. Deferoxamine increases urinary iron excretion and is the only chelator currently available for chronic administration. Daily administration of deferoxamine results in negative iron balance in most patients by the age of 10; this study was designed to determine whether the onset of cardiac complications was delayed and life prolonged by iron removal.

This trial began in 1978. Its forerunner was a study involving both deferoxamine and ascorbic acid. Although ascorbic acid promotes iron removal, its administration was followed by cardiac deterioration in several patients. In this study, patients receiving subcutaneous deferoxamine were randomized to receive either ascorbic acid or placebo, thereby providing a controlled test of this agent in treatment of iron overload. Sixty-five patients with homozygous beta-thalassemia participated in the long-term chelation trial. Of these, 49 were randomized to the ascorbic acid trial.

Several noninvasive techniques have been developed to evaluate organ function in iron-overloaded patients, thereby facilitating the assessment of chelation therapy. These techniques included chest x-rays, electrocardiograms, echocardiograms, and 24-hour Holter monitoring to assess cardiac function. Liver function was evaluated by standard liver function tests, CAT scan, and live biopsy. During the last six years of the study, hepatic iron stores were measured magnetically with a dual channel superconducting quantum-interference susceptomer. Endocrine function was also assessed by standard tests.

DESIGN NARRATIVE:

All patients received subcutaneous deferoxamine and iron removal was determined by measurement of serum ferritin and periodic non-invasive measurements of liver iron concentration. Clinical status was evaluated by non-invasive testing of cardiac and endocrine function.

The study completion date listed in this record was inferred from the last publication listed in the Citations section of this study record.

ELIGIBILITY:
Males and females, 5 years or older, with transfusional hemochromatosis.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1978-01; Study Completion 1994-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Young — Laboratory of Hematology, NHLBI

REFERENCES:
- [Background] Nienhuis AW, Griffith P, Strawczynski H, Henry W, Borer J, Leon M, Anderson WF. Evaluation of cardiac function in patients with thalassemia major. Ann N Y Acad Sci. 1980;344:384-96. doi: 10.1111/j.1749-6632.1980.tb33677.x. PMID 6930878
- [Background] Brittenham GM, Griffith PM, Nienhuis AW, McLaren CE, Young NS, Tucker EE, Allen CJ, Farrell DE, Harris JW. Efficacy of deferoxamine in preventing complications of iron overload in patients with thalassemia major. N Engl J Med. 1994 Sep 1;331(9):567-73. doi: 10.1056/NEJM199409013310902. PMID 8047080